CLINICAL TRIAL: NCT05638724
Title: Munich Long COVID Registry for Children, Adolescents, and Adults (MLC-R)
Brief Title: Munich Long COVID Registry for Children, Adolescents, and Adults
Acronym: MLC-R
Status: Recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Charite University, Berlin, Germany (Other); Ruhr University of Bochum, Germany (Unknown); Technical University of Dresden, Germany (Unknown); University of Freiburg (Other); University of Hamburg-Eppendorf (Other); Leipniz University Hannover, Germany. (Unknown); Saarland University Homburg,Germany. (Unknown); Friedrich Schiller University Jena, Germany (Unknown); University of Kassel, Germany. (Unknown); University of Cologne (Other)
Responsible Party: Sponsor
Other Study IDs: MLC-R Study
Record Dates: First submitted 2022-11-03; First posted 2022-12-06 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-12

CONDITIONS: Post-COVID Condition
Keywords: Long COVID; Post-COVID; ME/CFS; CFS/ME; SARS-CoV-2; COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The MLC-R aims to create a large-scale registry that provides data on epidemiology, phenotypes, and disease trajectories of and health care for Long COVID at any age in Germany, which can be used for future clinical trials.

DETAILED DESCRIPTION:
Infections with the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) have been observed in Germany since January 2020 and can result in acute coronavirus disease 2019 (COVID-19) as well as in long-term sequela, referred to as Long COVID. The umbrella term Long COVID comprises ongoing new SARS-CoV-2-associated symptoms later than four weeks from the onset of acute COVID-19. The term Post-COVID-Condition (PCC) was introduced by the WHO and stands for ongoing or new SARS-CoV-2-associated symptoms, which persisted for at least two months. These symptoms often include fatigue, brain fog, dyspnea, orthostatic intolerance, as well as exercise intolerance, with a worsening of symptoms after mild daily activities (post-exertional malaise, PEM). PCC can severely impair daily function, social participation, and health-related quality of life. The prevalence was estimated as up to 15% in infected people with pre-Omicron variants and lower with Omicron variants. Risk factors include female gender and pre-existing morbidity, with low risk in young children. The most severe form of PCC in people with initially mild or moderate COVID-19 is myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS). The prevalence of ME/CFS was shown to increase in the context of the pandemic. While progress has been made in deciphering the pathogenesis of acute COVID-19, the mechanisms of Long COVID/PCC are poorly understood. Increasing evidence indicates that remaining viral particles, as well as inflammation, altered microcirculation, dysfunction of the autonomic nervous system, and/or autoimmunity, may contribute.

With the web-based German MLC-R, we aim at deep phenotyping of PCC, identification of subtypes and risk factors, describing trajectories of the disease and patient journeys, and providing clinical data for future clinical trials. Patients are also invited to contribute biosamples for future translational research.

ELIGIBILITY:
Inclusion Criteria:

I. Written informed consent of the patient or legal guardian.

II. Confirmed SARS-CoV-2 vaccination and/or confirmed or probable SARS-CoV-2 infection: Positive SARS-CoV-2 polymerase chain reaction (PCR) or rapid antigen test (AST), documented probable COVID-19 (e.g., typical CT scan), probable COVID-19 with a history of high-risk contact, anti-SARS-CoV-2-N antibodies (and/or in non-vaccinated people -S-IgG antibodies) following probable COVID-19.

III. Additional ICD-10 codes: U09.9!V: Suspected post-COVID-19 condition, unspecified; U12.9!V: suspected adverse reactions to COVID-19 vaccine use, unspecified (post-COVIDvac condition).

Exclusion Criteria:

* Any subsequent medical data that question the diagnosis of PCC or post-COVIDvac condition
* Clinical picture can be explained by another underlying disease.
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with PCC
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2027-07-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
Phenotyping of Post-COVID condition: Medical History | 5 years
  Routine assessment of the medical history, such as current and previous medication, vaccinations, comorbidities, and more, to achieve a profound and detailed Post-COVID condition phenotype.
Phenotyping of Post-COVID condition: Physical Examination | 5 years
  Routine physical examination to achieve a profound and detailed Post-COVID condition phenotype.
Phenotyping of Post-COVID condition: Laboratory Parameters | 5 years
  Measurement of a routine set of laboratory parameters including blood tests (cell count, C-reactive protein, organ function, immunoglobulins, antibodies, etc.) and urine/stool analysis (calprotectin, blood) to achieve a profound Post-COVID condition phenotype.
Phenotyping of Post-COVID condition: Functional Tests | 5 years
  Technical exams (e.g. pulmonary function tests, electrocardiography, ultrasound, magnetic resonance imaging, etc.) will be performed as indicated to achieve a profound and detailed Post-COVID condition phenotype.

SECONDARY OUTCOMES:
Analyzation of numbers of physicians involved | 5 years
  Patients' journeys will be analyzed in terms of the number of physicians involved
Evaluation of kind of spezializations of physicians involved | 5 years
  Patients' journeys will be analyzed in terms of the kind of specializations of physicians involved
Evaluation of kind of the latency of symptoms | 5 years
  Patients' journeys will be analyzed in terms of the kind of specializations of physicians involved
Evaluation of kind of the onset of therapy | 5 years
  Patients' journeys will be analyzed in terms of the latency from symptom onset to initiation of therapy in months.
Definition of Sub-cohorts | 5 years
  Sub-cohorts are identified using routine data. By means of e.g. trigger, disease severity (e.g. Bell score from the worst outcome with 0 points till the best outcome with 100 points), daily functioning (e.g. SF-36).
Prevalence of Comorbidities | 5 years
  Prevalence of comorbidities of patients with Post-COVID condition will be analyzed.
Identification of Candidate Prognostic Markers | 5 years
  Correlation of routine clinical data (e.g., medical history, routine laboratory, and physical examination) with clinical outcome (e.g., health-related quality of life, disease severity, and social participation).

CONTACTS AND LOCATIONS:
Overall Officials: Uta Behrends, Prof. Dr. med., Principal Investigator — MRI Chronic Fatigue Center for Young People (MCFC), Children's Hospital, Technical University of Munich & Munich Municipal Hospital
Locations (1):
- MRI Chronic Fatigue Center for Young People (MCFC) Children's Hospital, Technical University of Munich & Munich Municipal Hospital, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided